CLINICAL TRIAL: NCT01773122
Title: Safety, Tolerability, and Pharmacokinetics of Dapsone in Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 225678-004
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dapsone Formulation A (Experimental): Dapsone Formulation A applied once daily to the face, upper chest, upper back, and shoulders for 28 days.
  Interventions: Drug: Dapsone Formulation A
- Dapsone Formulation B (Experimental): Dapsone Formulation B applied once daily to the face, upper chest, upper back, and shoulders for 28 days.
  Interventions: Drug: Dapsone Formulation B
- Dapsone Formulation C (Experimental): Dapsone Formulation C applied once daily to the face, upper chest, upper back, and shoulders for 28 days.
  Interventions: Drug: Dapsone Formulation C
- Dapsone 5% Gel (Active Comparator): Dapsone 5% gel (ACZONE®) applied twice daily to the face, upper chest, upper back, and shoulders for 28 days.
  Interventions: Drug: Dapsone 5% Gel

INTERVENTIONS:
Drug: Dapsone Formulation A — Dapsone Formulation A applied once daily to the face, upper chest, upper back, and shoulders for 28 days.
  Arms: Dapsone Formulation A
Drug: Dapsone Formulation B — Dapsone Formulation B applied once daily to the face, upper chest, upper back, and shoulders for 28 days.
  Arms: Dapsone Formulation B
Drug: Dapsone Formulation C — Dapsone Formulation C applied once daily to the face, upper chest, upper back, and shoulders for 28 days.
  Arms: Dapsone Formulation C
Drug: Dapsone 5% Gel — Dapsone 5% gel (ACZONE®) applied twice daily to the face, upper chest, upper back, and shoulders for 28 days.
  Other Names: ACZONE®
  Arms: Dapsone 5% Gel

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics (PK) of dapsone in subjects with acne vulgaris following 28 days of dosing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acne vulgaris
* Willing to avoid excessive or prolonged exposure to ultraviolet light (e.g., sunlight, tanning beds) throughout the study
* If male, the subject must agree to shave the facial treatment area and agree to maintain his routine shaving regimen for the duration of the study
* willing to avoid applying moisturizers, sunscreens, cosmetics (except eye and lip makeup), and chemical peels throughout the study

Exclusion Criteria:

* Oral acne treatments within 6 months

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2013-01-21 (Actual); Primary Completion 2013-05-05 (Actual); Study Completion 2013-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- College Station, Texas, United States

REFERENCES:
- [Background] Jarratt MT, Jones TM, Chang-Lin JE, Tong W, Berk DR, Lin V, Kaoukhov A. Safety and Pharmacokinetics of Once-Daily Dapsone Gel, 7.5% in Patients With Moderate Acne Vulgaris. J Drugs Dermatol. 2016 Oct 1;15(10):1250-1259. PMID 27741344

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol was amended mid-study to exclude patients <16 years.
Period: Overall Study
Arm/Group | Dapsone Formulation A | Dapsone Formulation B | Dapsone Formulation C | Dapsone 5% Gel
Started | 20 | 19 | 19 | 19
Completed | 17 | 18 | 19 | 18
Not Completed | 3 | 1 | 0 | 1
Not completed — Due to amended age eligibility criteria | 3 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapsone Formulation A | Dapsone Formulation B | Dapsone Formulation C | Dapsone 5% Gel | Total
Number analyzed (Participants) | 20 | 19 | 19 | 19 | 77
Age, Customized [Number; unit: Participants]
  12 to 17 years | 8 | 7 | 7 | 7 | 29
  18 to 35 years | 12 | 12 | 12 | 12 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 10 | 9 | 36
  Male | 12 | 10 | 9 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Level (Cmax) of Dapsone
Description: Cmax is the maximum plasma level following multiple doses of dapsone. Plasma is the liquid component of the blood in which the blood cells are suspended.
Time Frame: Day 28
Population: All treated subjects with data for this time point
Measure: Mean (Standard Deviation); unit: Nanograms/Milliliter (ng/mL)
Arm/Group | Dapsone Formulation A | Dapsone Formulation B | Dapsone Formulation C | Dapsone 5% Gel
Number analyzed (Participants) | 17 | 18 | 19 | 18
Nanograms/Milliliter (ng/mL) | 11.7 (5.5) | 14.1 (8.8) | 13.0 (6.8) | 17.6 (6.7)

2. Secondary Outcome: Maximum Plasma Level (Cmax) of Dapsone Metabolites
Description: Cmax is the maximum plasma level following multiple doses of dapsone. Plasma is the liquid component of the blood in which the blood cells are suspended. The dapsone metabolites are N-acetyl dapsone and dapsone hydroxylamine.
Time Frame: Day 28
Population: All treated subjects with data for this time point
Measure: Mean (Standard Deviation); unit: Nanograms/Milliliter (ng/mL)
Arm/Group | Dapsone Formulation A | Dapsone Formulation B | Dapsone Formulation C | Dapsone 5% Gel
Number analyzed (Participants) | 17 | 18 | 19 | 18
Nanograms/Milliliter (ng/mL)
  N-Acetyl Dapsone | 5.44 (4.25) | 6.00 (3.85) | 6.47 (5.43) | 11.7 (8.8)
  Dapsone Hydroxylamine | 0.908 (0.433) | 1.11 (0.46) | 1.19 (0.76) | 1.47 (0.56)

ADVERSE EVENTS:
Description: The Safety Population consisted of all subjects who received at least 1 dose of study medication. The Safety Population was used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | Dapsone Formulation A | Dapsone Formulation B | Dapsone Formulation C | Dapsone 5% Gel
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 20/20 | 16/19 | 10/19 | 11/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dapsone Formulation A (N=20) | Dapsone Formulation B (N=19) | Dapsone Formulation C (N=19) | Dapsone 5% Gel (N=19)
Headache (Nervous system disorders) | 6 | 2 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1/8 | 2/9 | 0/10 | 1/9
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Medical Device Pain (General disorders) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Tinea Versicolour (Infections and infestations) | 1 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.